CLINICAL TRIAL: NCT02010281
Title: Long-term Efficacy of Repetitive Transcranial Magnetic Stimulation (rTMS) of the Motor or Prefrontal Cortex in Peripheral Neuropathic Pain: a Multicenter Randomized Placebo Controlled Trial
Brief Title: Analgesic Effects of rTMS in Peripheral Neuropathic Pain
Acronym: TRANSNEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P120126; AOM 120141 (Other: APHP)
Record Dates: First submitted 2013-11-07; First posted 2013-12-12 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Neuropathic Pain
Keywords: rTMS; peripheral neuropathic pain; randomized controlled trial
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- rTMS of the motor cortex (Magventure) (Experimental): experimental : rTMS of the motor cortex : repetitive magnetic stimulation targeting the motor cortex assisted by neuronavigation
  Interventions: Device: rTMS of prefrontal or motor cortex
- rTMS placebo (magventure) (Placebo Comparator): sham stimulation of the motor or prefrontal cortex with the placebo face of the device
  Interventions: Device: rTMS of prefrontal or motor cortex
- rTMS prefrontal cortex (magventure) (Experimental): Experimental : repetitive transcranial stimulation targeting the prefrontal cortex as indicated by neuronavigation
  Interventions: Device: rTMS of prefrontal or motor cortex

INTERVENTIONS:
Device: rTMS of prefrontal or motor cortex — description:rTMS of the motor or prefrontal cortex (repetitive magnetic stimulation targeting the motor or prefrontal cortex) assisted with neuronavigation

SUMMARY:
This study aims to evaluate the long term efficacy over 25 weeks of repeated sessions of magnetic transcranial stimulation of the motor cortex or prefrontal cortex on average pain intensity, quality of life, sleep, neuropathic symptoms, return to work, in patients with peripheral neuropathic pain.

The medical device of study: transcranial magnetic stimulator (TMS).

DETAILED DESCRIPTION:
The present multicenter parallel session randomized placebo controlled study (4 French centers) aims to evaluate the long term efficacy over 25 weeks of repeated sessions of magnetic transcranial stimulation of the motor cortex or prefrontal cortex on average pain intensity (primary outcome) and several secondary outcome measures (e.g. quality of life, sleep, neuropathic symptoms, return to work), in patients with peripheral neuropathic pain.

The patients will be randomized to receive one of 3 treatment arms : rTMS of the motor cortex, rTMS of the prefrontal cortex, or placebo (sham stimulation) of the motor or prefrontal cortex. The study will be double blind, eg the patient and the investigator will not know the nature of treatment. the stimulation protocol will consist of an induction phasse of 5 daily sessions then a maintenance phase of several sessions : 3 sessions a week apart, 3 sessions a fortnight apart, and 3 sessions 3 weeks apart. The statistical analysis will be conducted in the intent to treat population and using a modified ITT analysis excluding all the patients with protocol violation (primary outcome). The per protocol population will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Peripheral neuropathic pain (unilateral or bilateral) probable or defined according to the criteria proposed in 2008 (Treede et al 2008),
2. Diagnostic DN4 questionnaire score greater than or equal to 4/10 (Bouhassira et al 2005),
3. chronic pain, the average intensity is greater than or equal to 40/100
4. Daily or almost daily pain (at least 4 days out of 7)
5. This pain is present for more than 6 months
6. Patients over 18 and under 75 years old
7. Patients who signed informed consent,
8. Patients whose pain medication is stable for 15 days before inclusion, and will not need to be changed during the study period,
9. Patients who can be monitored during the study period (30 weeks)
10. Patients insured by a health insurance plan or entitled.

Exclusion Criteria:

1. Previous treatment using rTMS,
2. Work Accident or dispute
3. rTMS Cons-indications (ECT treatment during the previous month, epilepsy and / or a history of epilepsy; history of head trauma, neurosurgical lesion, intracranial hypertension, metal clip, pacemaker, pregnant or lactating women)
4. Abuse of drugs or psychoactive substances (DSM IV)
5. Central neuropathic pain,
6. Neuropathic pain within the framework of a progressive disease (HIV, cancer, non-stabilized system disease)
7. Neuropathic pain very limited extent, of neuroma type
8. Current major depression or psychosis according to DSM IV criteria,
9. Intermittent pain,
10. Pain for less than six months,
11. Presence of another pain more severe than the one justifying the inclusion
12. Lack of proper filling of self-assessment of pain from baseline and randomization (at least 4 weekly pain scores 7 days) notebooks
13. Lack of stability of pain scores on two successive evaluations, defined as a change of more than 30% between the two assessments of the average pain on the short questionnaire about pain between the first two visits inclusion
14. Subject unable to understand informed consent, under guardianship,
15. Subject who refuses to stop or can not stop prohibited treatment during the study,
16. Patients participating in another research protocol involving a drug within 30 days before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2019-05-11 (Actual)

PRIMARY OUTCOMES:
Change in average pain intensity from baseline to week 25 | each visit for up to 25 weeks
  Change in average pain intensity from baseline to week 25, average pain intensity corresponds to average pain over the last 24 hours on the Brief Pain Inventory

SECONDARY OUTCOMES:
change in minimal pain intensity over the last 24 hours from baseline to week 25 | each visit for up 25 weeks
  change in minimal pain over the last 24 hours on the Brief Pain inventory
quality of life assessment | each visit up to 25 weeks
  quality of life on the Eurogol questionnaire
Proportion of responders to rTMS | at the end of treatment (25 weeks)
  Proportion of responders (patients whose pain is improved by at least 30% and 50% compared to their pain before treatment
Predictors of the response | Baseline
  Evaluation of predictors of response (nature of neuropathic symptoms, severity of anxiety or depressive symptoms, presence or absence of mechanical allodynia, or dramatization importance of catastrophism related to pain)
Safety evaluation | each follow up visit for up to 25 weeks
  Collection of side effects at each session and between sessions of rTMS
Onset of the analgesic effect of rTMS | one mont afer the beginning of rTMS
  Determine the onset of the analgesic effect based on patient pain diaries for up to 1 month
Return to work | 25 weeks
  Return to work on a specific questionnaire at the end of the study
Maximal pain | each visit up to 25 weeks
  Maximal pain over the past 24 hours on the Brief Pain Inventory
Pain right now | each visit up to 25 weeks
  Pain right now immediately after each rtMS session and between sessions for up to 25 weeks
Sleep | each visit up to 25 weeks
  sleep quality and quantity on MOS sleep
Neuropathic symptoms | each visit up to 25 weeks
  Neuropathic symptoms on the Neuropathic Pain Symptom Inventory

CONTACTS AND LOCATIONS:
Overall Officials: NADINE ATTAL, MD, PhD, Principal Investigator — Pain evaluation and treatment center, CHU A Paré, 92104 Boulogne Billancourt, France
Locations (1):
- Pain evaluation and treatement center, CHU Ambroise Paré, Boulogne-Billancourt, Hauts-de-Seine, France

REFERENCES:
- [Derived] Attal N, Branders S, Pereira A, Bouhassira D. Prediction of the response to repetitive transcranial magnetic stimulation of the motor cortex in peripheral neuropathic pain and validation of a new algorithm. Pain. 2025 Jan 1;166(1):34-41. doi: 10.1097/j.pain.0000000000003297. Epub 2024 Jun 14. PMID 38875120
- [Derived] Attal N, Poindessous-Jazat F, De Chauvigny E, Quesada C, Mhalla A, Ayache SS, Fermanian C, Nizard J, Peyron R, Lefaucheur JP, Bouhassira D. Repetitive transcranial magnetic stimulation for neuropathic pain: a randomized multicentre sham-controlled trial. Brain. 2021 Dec 16;144(11):3328-3339. doi: 10.1093/brain/awab208. PMID 34196698